CLINICAL TRIAL: NCT01593839
Title: Functioning Disturbance in Chronic Back Pain: Altered Muscle Metabolism
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: The Research Council of Norway (Other)
Responsible Party: Sponsor
Other Study IDs: 182006/V50; 08/5253 Personvernombudet RRHF
Record Dates: First submitted 2012-05-04; First posted 2012-05-08 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-05

CONDITIONS: Chronic Non-specific Low Back Pian

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Interstitial
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The main objective of this study is to investigate the muscle metabolism in individuals with chronic non-specific low back pain (CNSLBP) to enhance our understanding of chronic back pain.

ELIGIBILITY:
The NSCBP group:

* At least 6 patients will be included in this study.
* All patients referred to Vestfold Hospital Trust, Kysthospitalet, diagnosed with chronic NSCBP >3 months duration will be invited to participate in the study. The invitation will be in a written form.

Exclusion Criteria:

* anamnesis of medical or drug abuse,
* surgery on the musculoskeletal system of the trunk,
* known congenital malformation of the spine or scoliosis,
* body mass index > 27 kg/m2,
* systemic-neurological-degenerative disease,
* history of stroke,
* psychiatric disorder,
* pregnancy and abnormal blood pressure. The subjects will be asked not to use any medications except for paracetamol preparations one week before examination and instructed not to perform any back-straining exercise for 48 h prior to the study, except for ordinary daily working and/or leisure activities.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Persons referred to Hospital of rehabilitation due to chronic non-specific low back pain
Sampling Method: Non-Probability Sample
Enrollment: 6 (Estimated)
Dates: Start 2012-05; Primary Completion 2013-06 (Estimated); Study Completion 2013-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Kysthospitalet, Vestfold Hospital Trust, Stavern, Norway